CLINICAL TRIAL: NCT01532258
Title: Effectiveness of an Eight Week Online Mediterranean Based Diet in an Overweight or Obese Outpatient Primary Care Population
Brief Title: Effectiveness of an Eight Week Online Mediterranean Based Diet
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Online program required re-design
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Linda Libertini, Research Coordinator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB# 11-475
Record Dates: First submitted 2011-09-23; First posted 2012-02-14 (Estimated); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Obesity
Keywords: BMI; Weight loss; Nutrition; Diet; Mediterranean diet; Online program; web-based program; Oxidative stress; F2 isoprostanes
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Group (No Intervention): No intervention provided. These participants will receive access to the Go! Foods for You program after the research trial has been completed (12 weeks after registration).
- GFFY-1 without weekly MA support (Active Comparator): Utilization of the 8-week online nutrition program Go! Foods for You without weekly contact from staff at the medical provider's office.
  Interventions: Behavioral: Go! Foods for You without Weekly MA Support.
- GFFY-2 with weekly MA support (Active Comparator): Utilization of the 8-week online nutrition program combined with weekly contact from the staff at the medical provider's office.
  Interventions: Behavioral: Go! Foods for You with Weekly MA Support.

INTERVENTIONS:
Behavioral: Go! Foods for You without Weekly MA Support. — * Participants access and utilize an 8-week online program which provides educational materials and weekly activities based on a Mediterranean diet and dietary "practices" that have been associated with healthy weights.
  * Each day participants receive educational materials related to the nutritional science of a Mediterranean diet. Each week (1) a new theme for the daily educational materials is presented and (2) participants are asked to schedule "activities" on a built in calendar and practice the activity throughout the week.
  Arms: GFFY-1 without weekly MA support
Behavioral: Go! Foods for You with Weekly MA Support. — * Participants access and utilize an 8-week online program which provides educational materials and weekly activities based on a Mediterranean diet and dietary "practices" that have been associated with healthy weights.
  * In addition to the 8-week online program, participants receive weekly support by Medical Assistants (MA) over the phone or by email to establish a relationship and maintain program adherence by discussing the previous week's behavioral goals and setting weekly behavioral goals.
  Arms: GFFY-2 with weekly MA support

SUMMARY:
This research is examining whether an 8-week online nutritional programming based on a Mediterranean diet can achieve meaningful increase intake of a Mediterranean based diet and improvements in measures of body weight and laboratory measures of oxidative stress, a risk marker for cardiovascular disease. This study will also examine whether weekly short support and communication from a medical assistant (MA) in a primary care setting in addition to the online program will result in better program adherence and have a positive impact on health.

DETAILED DESCRIPTION:
Eligible participants will be identified by primary care providers or their staff at clinical outpatient site(s). Study is 3-arm randomized control trial where participants will be randomized to 1) Control group (CTL)-will not receive access to online program nor intervention for first 12 weeks; 2) GFFY-1-will receive access to online program without MA intervention 3) GFFY-2-will receive access to online program and MA intervention with weekly phone call. The core of the intervention is an 8-week Mediterranean diet and behavioral online program called "Go! Foods for You (GFFY)" which is offered on the Cleveland Clinic's 360.5.com website. The research will last for 24 weeks. Questionnaire data and biometric measurements will be collected at pre and post intervention (0-8 weeks) and at followup (12 and 24 weeks). Regardless of randomization, participants will be asked to provide their weight every week and an activity log at the end of each week of the program. A urine sample to measure F2-isoprostane will be collected at week 0 and 12 for GFFY-2 and CTL groups.

A preparatory phase requiring the involvement of MAs to provide weekly support to participants is necessary to test process and communication with MAs. Enrollment of 10-20 volunteers for the preparatory phase is desired. Data collected during this phase will not be part of study analysis. To test data collection process, we may ask a few participants to complete baseline questionnaire only.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 25 or greater.
* Age 18 to 70 years old.
* Patient of a participating Internal Medicine or Family Medicine primary care provider at a Cleveland Clinic Family Health Center.
* Registered on the Cleveland Clinic's electric medical records, My Chart.

Exclusion Criteria:

* Women who are pregnant or planning to be pregnant in the next 6 months.
* No easy internet and email access at place of residence.
* No access to a scale at place of residence for weekly weight measurement.
* Sudden unintentional weight loss or weight gain in the past 3 months due to medical illness
* Currently involved in a weight loss program
* unwilling to be in the wait-list control group where participant will not have access to the program for 3 months
* unwilling to log onto the internet on a regular basis for the duration of the study (3-4 months)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 12 weeks
  To see if the 8-week Mediterranean diet online program (GFFY) can lead to weight loss at 12 week.
Effect of Weekly Communications on Adherence and Program Efficacy | 12 weeks
  To see if extension of the patient/medical provider relationship through weekly emails by a medical assistant who addresses the program behavioral goals set by the patient leads to greater weight loss.

SECONDARY OUTCOMES:
Effect on Oxidative Stress | 12 weeks
  To see if the program reduces bio markers of oxidative stress (F2 isoprostanes) for participants in the GFFY-2 compared to the CTL group.
Correlation between MA Support and Program Utilization | 12 weeks
  To see if participation in GFFY with MA support can improve program participation as measured by 8-week program completion rate and average weekly activities completed during the 8-week program.
Effect on Physical and Mental Health | 12 weeks
  To see if an 8-week Mediterranean diet online program help improve overall physical and mental health as measured by the RAND Corporation Health Survey tool (SF36Rand).
Sustainability of Weight Loss | 24 weeks
  To see if weight loss from participation in the GFFY programs is sustained at 24 weeks (6 months) follow-up.
Dietary Improvements | 12 weeks
  To see if participation in GFFY increases fiber intake, percentage fat and fruit and vegetable consumption as measured by a brief online food screening questionnaire
Increase in Intake of a Mediterranean-based Diet | 12 weeks
  To see if participation in GFFY increases intake of a Mediterranean based diet as measured by a short Mediterranean diet questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States